CLINICAL TRIAL: NCT04874129
Title: Phase 1 to Evaluate the Safety and Pharmacokinetic Characteristics of Fixed-dose Combination of YYC506
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YYPCT_YYC506_102
Record Dates: First submitted 2021-04-20; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Intervention Model Description: ramdomized, open-label, single-dose, two-way crossover study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Group (Other): Two-way Crossover
  Interventions: Drug: YYC506-T and YYC506-A (phase 1); Drug: YYC506 (phase 2)
- B Group (Other): Two-way Crossover
  Interventions: Drug: YYC506 (phase 1); Drug: YYC506-T and YYC506-A (phase 2)

INTERVENTIONS:
Drug: YYC506-T and YYC506-A (phase 1) — Comparator
  Other Names: Comparator
  Arms: A Group
Drug: YYC506 (phase 1) — Test
  Other Names: Test
  Arms: B Group
Drug: YYC506-T and YYC506-A (phase 2) — Comparator
  Other Names: Comparator
  Arms: B Group
Drug: YYC506 (phase 2) — Test
  Other Names: Test
  Arms: A Group

SUMMARY:
To evaluate the safety and pharmacokinetics characteristics between YYC506 and concomitant administration of YYC506-T and YYC506-A

DETAILED DESCRIPTION:
Phase 1 to evaluate the safety and pharmacokinetics characteristics between YYC506 and concomitant administration of YYC506-T and YYC506-A. Which is designed as ramdomized, oral, single dose, two-way crossover.

ELIGIBILITY:
Inclusion Criteria:

* Over 19 ages healthy men
* Over 50.0kg, 18.0kg/m2 ≤ BMI ≤ 30.0kg/m2
* Men who don't have congenital disease and other cronic disease need to be cared. etc.

Exclusion Criteria:

* Men who have congenital liver disease (AST, ALT, CK ≥ 2X ULN)
* Men who have drunken or eatten something including caffeine within 24 hours before. etc.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters: Cmax | Until 48 hours
  Cmax
Pharmacokinetic parameters: AUC | Until 48 hours
  YYC506-T, YYC506-A, YYC506 AUC

CONTACTS AND LOCATIONS:
Overall Officials: Min Kyu Park, PhD, Study Chair — Chungbuk National University Hosipital.
Locations (1):
- Chungbuk National Unviersity Hosipital, Cheongju-si, South Korea

IPD SHARING:
Plan to Share IPD: No